CLINICAL TRIAL: NCT05364255
Title: A Phase I, Open-Label, Single-Dose, Single-Period Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]AZD9833 After Oral Administration in Healthy Post-Menopausal Female Subjects
Brief Title: A Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]AZD9833
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8532C00005; 2022-000834-40 (EudraCT Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: ER-positive, HER2-negative Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]AZD9833 (D8532C00005) (Experimental): Oral Solution, 75 mg (NMT 0.67 MBq)
  Interventions: Drug: [14C]AZD9833 Oral Solution, 75 mg

INTERVENTIONS:
Drug: [14C]AZD9833 Oral Solution, 75 mg — Oral Solution, 75 mg (NMT 0.67 MBq) - oral, fasted

SUMMARY:
The Sponsor is developing the test medicine, AZD9833 for the potential treatment of estrogen receptor (ER)-positive breast cancer.

This single-part, healthy volunteer study will try to identify how the test medicine is taken up, broken down and removed from the body. To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14) which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

This study will take place at one non-NHS site, and will consist of a single study period involving up to 6 post-menopausal female volunteers, aged between 50 to 70 years.

DETAILED DESCRIPTION:
The Sponsor is developing the test medicine, AZD9833 for the potential treatment of estrogen receptor (ER)-positive breast cancer.

Breast cancer is the second most common type of cancer in the UK and worldwide. Most women diagnosed with breast cancer are over the age of 50, but younger women and men can also get breast cancer. AZD9833 has the potential to prevent ER activity and increase overall survival in advanced breast cancer patients.

This single-part, healthy volunteer study will try to identify how the test medicine is taken up, broken down and removed from the body. To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14) which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

This study will take place at one non-NHS site, and will consist of a single study period involving up to 6 post-menopausal female volunteers, aged between 50 to 70 years.

On Day 1, volunteers will receive a 75 mg dose of [14C]AZD9833 oral solution in the fasted state (on an empty stomach).

Volunteer's blood, urine and faeces will be taken throughout the study for analysis of the test medicine and it's breakdown products (metabolites) and for volunteer safety.

Volunteers will remain in the clinical unit until Day 8, however if the relevant radioactivity criteria have not been met, volunteers may be required to remain at the clinic until Day 10. If relevant criteria have not been met at this point, home collections of urine and/or faeces may be required.

Volunteers are expected to be involved in this study for approximately 6 weeks from screening to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Aged between 50 to 70 years inclusive at the time of signing informed consent
* Healthy post-menopausal females, defined as post-menopausal by fulfilling the following criterion:

  (a) amenorrhoea for at least 12 months following cessation of all exogenous hormonal treatments and without an alternative medical or surgical cause and confirmed by an FSH result of ≥30 IU/L
* Must be willing and able to communicate and participate in the whole study
* Have a body mass index (BMI) between 19.0 to 35.0 kg/m2, weigh at least 50 kg and no more than 100 kg inclusive as measured at screening.
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP
* History of or ongoing clinically significant visual disturbances including but not limited to visual hallucinations, migraine with visual symptoms, blurred vision, frequent floaters/flashes associated with other symptoms such as dizziness
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, at screening as judged by the Investigator
* Any clinically significant abnormal findings in vital signs at screening as judged by the Investigator, including systolic BP <100 mmHg, diastolic BP <50 mmHg or heart rate <50 bpm. Vital signs outside these limits can be repeated once for confirmation
* Any clinically significant abnormalities on 12-lead ECG at screening, as judged by the Investigator, including non-sinus rhythms, PR interval <120 msec or >220 msec, ventricular rate <50 bpm or >100 bpm, QRS interval >120 msec, or QTcF >470 msec as a mean of triplicate. ECGs can be repeated once in triplicate if parameters are outside these limits for confirmation
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <60 mL/min/1.73m2 using the Cockcroft-Gault equation
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), and human immunodeficiency virus (HIV) 1 and 2 antibodies
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 4 weeks prior to Day 1, or less than 5 elimination half-lives + 6 days prior to Day 1, whichever is longer. Note: subjects consented and screened, but not administered IMP in this study or a previous Phase I study, are not excluded
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9833. Hay fever is allowed unless it is active
* Any known or suspected hypersensitivity or contraindication to the components of the study drug, AZD9833, judged to be clinically relevant by the investigator
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Positive screen for drugs of abuse at screening or on each admission to the study centre
* Regular alcohol consumption >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
* A confirmed positive alcohol breath test at screening or admission
* Subjects who are taking, or have taken:

  1. any prescribed or over-the-counter drug (other than up to 4 g of paracetamol per day ) or herbal remedies in the 14 days before IMP administration or longer if the medication has a long half-life. COVID-19 vaccines are accepted concomitant medications. Exceptions may apply, as determined by the Investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no PD activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study
  2. atropine or atropine containing drugs, in the 14 days before IMP administration
  3. Systemic oestrogen-containing hormone replacement therapy in the 6 months prior to IMP administration
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks or 5 half-lives (whichever is longer) or any drugs with a known risk, potential risk or conditional risk for QTca prolongation as defined and outlined in the Credible Meds website within 4 weeks prior to Day 1
* Subjects who do not agree to avoid the to use warfarin or phenytoin (and other coumarin-derived vitamin K antagonist anticoagulants) for 2 weeks after administration of IMP
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g., >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the clinical unit
* Involvement of any Astra Zeneca, Quotient or study site employee or their close relatives
* Subjects who report to have previously received AZD9833 in the last 12 months
* Judgment by the Investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements
* Evidence of current SARS-CoV-2 infection
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator or delegate at screening
* Subjects with an anticipated need for major surgery and/or any surgery requiring general anaesthesia during the participation in the study (which may entail administration of atropine in an anaesthetic context)
* Failure to satisfy the Investigator of fitness to participate for any other reason

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The cumulative amount of AZD9833 excreted (CumAe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD9833 excreted
The cumulative amount of AZD9833 excreted, expressed as a percentage of the radioactive dose administered (Cum%Ae) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, expressed as a percentage, by measuring the cumulative amount of AZD9833 excreted
Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Plasma samples collected from pre-dose until 168 hours post-dose
  Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Urine samples collected from pre-dose until 168 hours post-dose
  Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Faeces samples collected from pre-dose until 168 hours post-dose
  Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry

SECONDARY OUTCOMES:
The amount of total radioactivity eliminated in urine (Ae) | Urine samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, by measuring the amount of AZD9833 excreted in urine by interval
The amount of total radioactivity eliminated in urine expressed as a percentage of the radioactive dose administered (%Ae) | Urine samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, expressed as a percentage, by measuring the amount of AZD9833 excreted in urine by interval
The cumulative amount of AZD9833 excreted in urine (CumAe) | Urine samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD9833 excreted in faeces.
The cumulative amount of AZD9833 excreted in urine, expressed as a percentage of the radioactive dose administered (Cum%Ae) | Urine samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, expressed as a percentage, by measuring the cumulative amount of AZD9833 excreted in urine
The amount of total radioactivity eliminated in faeces (Ae) | Faeces samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, by measuring the amount of AZD9833 excreted in faeces by interval
The amount of total radioactivity eliminated in faeces expressed as a percentage of the radioactive dose administered (%Ae) | Faeces samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, expressed as a percentage, by measuring the amount of AZD9833 excreted in faeces by interval
The cumulative amount of AZD9833 excreted in faeces (CumAe) | Faeces samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD9833 excreted in faeces.
The cumulative amount of AZD9833 excreted in faeces, expressed as a percentage of the radioactive dose administered (Cum%Ae) | Faeces samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity, expressed as a percentage, by measuring the cumulative amount of AZD9833 excreted in faeces
Time to maximum concentration (tmax) for AZD9833 and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the time to maximum concentration (tmax)
Maximum observed concentration (cmax) for AZD9833 and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the maximum observed concentration (cmax)
Area under the curve from time 0 to the time of last measurable concentration for AZD9833 and total radioactivity (AUC0-t) | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the area under the curve from time 0 to the time of last measurable concentration
Area under the curve from time 0 extrapolated to infinity for AZD9833 and total radioactivity (AUC0-inf) | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the area under the curve from time 0 extrapolated to infinity
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC%extr) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity
Terminal elimination half-life for AZD9833 (t1/2) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the terminal elimination half-life
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD9833 (λz) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the First order rate constant associated with the terminal (log-linear) portion of the curve
Total body clearance calculated after a single extravascular administration for AZD9833 (CL/F) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the total body clearance calculated after a single extravascular administration
Apparent volume of distribution based on the terminal phase for AZD9833 (Vz/F) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the apparent volume of distribution based on the terminal phase
Renal clearance for AZD9833 (CLr) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD9833 and total radioactivity by measuring the renal clearance
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Collection of blood samples until 168 hours post dose
  Assessment of total radioactivity in whole blood and plasma
Number of AE's experienced by subjects | AEs recorded from the time of informed consent until the follow up visit (approx 6 weeks)
  Safety and tolerability assessed through the incidence of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8532C00005&attachmentIdentifier=4f0f3eab-bcc6-4c2b-ada0-f36eb4127412&fileName=d8532c00005-study-synopsis_Redacted.pdf&versionIdentifier=